CLINICAL TRIAL: NCT07385196
Title: Trying to Define Ileorectal Syndrome: a Prospective Observational Study
Brief Title: Defining Ileorectal Syndrome: a Prospective Observational Study
Acronym: DEFINE-IRS
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozcem Ofkeli, operator doctor, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 828 - 19.12.2025
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Total Colectomy; Diarrhea; Urgency Incontinence; Soilings, Fecal
MeSH Terms: conditions — Diarrhea; Fecal Incontinence | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: survey study — The syndrome will be defined based on both patient observations and survey results.

SUMMARY:
1. Study Title: Trying to Define Ilorectal Syndrome: A Prospective Observational Study
2. Study Objective and Significance:

   Primary Objective:

   To prospectively evaluate the frequency, symptom severity, and impact on quality of life of ileorectal syndrome developing in patients who have undergone total colectomy and ileorectal anastomosis.

   Secondary Objectives:
   * To examine the relationship between postoperative bowel dysfunction and quality of life
   * To investigate clinical factors affecting symptom severity This study aims to contribute to postoperative follow-up and management strategies by revealing patient-centered outcomes of ileorectal syndrome.
3. Expected Benefits and Risks of the Study:

   Expected Benefits
   * Prospective and systematic evaluation of ileorectal syndrome
   * Identification of factors affecting the quality of life of these patients
   * Increased awareness in clinical follow-up Potential Risks
   * The study is observational and questionnaire-based and does not involve additional medical risks
   * No invasive procedures will be performed on the patients
4. Type, scope, and design of the planned study:

   * Type: Prospective, observational
   * Scope: Single-center
   * Design: Questionnaire-based clinical trial
5. Number of patients and volunteers to be included in the study, their qualifications, and the rationale for selection:

   * Total number of patients: 30
   * Age range: ≥18 years
   * Gender: Female and male This number was determined based on the appropriate patient population followed in our center.
6. Parameters to be examined:

   Demographic data (age, gender, BMI) Surgical indication Whether the surgery was performed openly or laparoscopically Level of anastomosis Maximum daily bowel movement frequency and duration Feeling of urgency Nocturnal bowel movements Fluid/gas incontinence - soiling Ileus in ADBG Whether electrolyte abnormalities developed Length of hospital stay Need for re-hospitalization Severity of symptoms based on patient reports and questionnaire questions
7. Where and by whom the parameters will be examined

   Data will be collected by the responsible investigator at the relevant clinic.
8. Which parameters to be used in the study are routine for that disease group and which are specific to the study?

   Routine: Demographic data, surgical information, laboratory results Study-Specific: Postoperative bowel functionality, symptom questionnaire
9. Estimated study duration, start and end dates:

   Start date: 1/1/2026 End date: 31/12/2026 Total duration: 12 months
10. Inclusion, exclusion, and withdrawal criteria:

    Inclusion Criteria
    * Having undergone total colectomy and ileorectal anastomosis
    * 18 years of age and older
    * Providing written informed consent Exclusion Criteria
    * Serious neurological disease affecting bowel function
    * Patients with incomplete follow-up data Withdrawal
    * At the patient's request
    * If follow-up cannot be completed
11. Termination criteria:

    By the ethics committee Termination decision Unforeseen circumstances preventing the conduct of the study
12. Statistical methods to be used in the evaluation of the data to be obtained as a result of the research:

    * Descriptive statistics (mean, median, percentage)
    * Parametric and non-parametric tests
    * Analysis of the relationship between symptom severity and quality of life
    * p < 0.05 statistical significance level

ELIGIBILITY:
Inclusion Criteria: Age ≥18 years

History of ileorectal anastomosis or preserved rectum following colorectal surgery

Ability to understand the study procedures and provide written informed consent

Willingness to participate in prospective follow-up assessments -

Exclusion Criteria:

Age <18 years

Permanent stoma

Total rectal excision

Inability to complete follow-up assessments

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with a history of ileorectal anastomosis and preserved rectum following colorectal surgery will be prospectively enrolled. The study population includes patients with or without bowel dysfunction symptoms suggestive of ileorectal syndrome. Participants will be followed prospectively to assess the prevalence and severity of bowel function-related symptoms over time.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence and severity of ileorectal syndrome-related bowel dysfunction symptoms assessed prospectively | Baseline and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- general surgery clinic(Gazi Yaşargil Tr and Res Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No